CLINICAL TRIAL: NCT03293823
Title: HARP-Project 1 Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Vankee Lin, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSRB00067540
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Aging; Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: 6-week cognitive training group vs. an active control group
Who Masked: Participant
Masking Description: Participants will not be informed whether it is an intervention or control group; instead they will be informed they will receive a computerized cognitive intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vision-based speed of processing (VSOP) cognitive training (Experimental): use the INSIGHT online program (Posit Science), which includes five training paradigms (Eye for detail, Peripheral challenge, Visual sweep, Double decision, Target tracker) that practice processing speed and attention. All exercises share visual components and focus on accuracy and fast reaction times. Participants respond either by identifying what object they see or where they see it on the screen. The training will automatically adjust the difficulty of each task based on the participant's performance, ensuring that the participants always operate near their optimal capacity. The training programs will automatically record the percentage of completion of each game and scores.
  Interventions: Behavioral: VSOP training
- active control (Active Comparator): The standardized computerized leisure activities program - MLA, including crossword puzzle, Sudoku, etc. will be used
  Interventions: Behavioral: MLA control

INTERVENTIONS:
Behavioral: VSOP training — a computerized cognitive training of attention and processing speed
  Arms: vision-based speed of processing (VSOP) cognitive training
Behavioral: MLA control — a computerized cognitive intervention of multiple mental leisure activities
  Arms: active control

SUMMARY:
Emerging evidence from social neuroscience suggests that prefrontal cortex (PFC), insular and anterior cingulate cortex (ACC) regulate social and emotional responses to acute threats to social connectedness among young adults. Deficient neural reserve or overused neural compensation resulting from neurodegeneration is commonly observed in these frontal regions in old age. This aging-related "neural depletion" may have implications for how older adults respond to social threats, potentially increasing maladaptive emotional and social behavioral responses, such as social anxiety and social avoidance, which contribute to social disconnectedness. The central hypothesis is that cognitive deficits and associated aging-related 'neural depletion' in the frontal regions will contribute to maladaptive social-emotional responses to a social stressor -- social exclusion. Ultimately, maladaptive responses to acute social stress, such as social anxiety and avoidance, can compromise social connectedness by increasing social strain and isolation. The investigators have recently developed a neuroplasticity-based cognitive training program, called vision-based speed of processing (VSOP) training, targeting multiple aspects of cognitive capacity (e.g., attention, working memory and inhibition) and incorporating the speed component to improve the efficiency of these cognitive processes. VSOP training also targets several neural networks seeded in ACC and insular (default mode network) or PFC (the frontal-striatal network and central executive network). These networks also overlap with neural substrates of emotion regulation. Notably, VSOP training appears to improve emotion regulation, as depressive symptoms were reduced in older adults following VSOP training. Finally, the autonomic nervous system (ANS), critical to stress adaptation, is regulated by these frontal regions. The objective of the proposed pilot study is to provide proof-of-concept for the hypothesis that improvements in older adults' cognitive capacity, frontal regions' neural efficiency, and ANS function via the VSOP training will be associated with more adaptive social-emotional response to social exclusion, which, in turn, should confer longer-term protection for older adults' sense of social connectedness. Randomized Controlled Trial Design: 30 older adults will be randomly assigned to engage in 6-week VSOP training, or to an active control group. Differential changes from baseline to post-training in cognitive capacity, neural efficiency, and ANS function, and sense of social connectedness, will be compared between VSOP control groups. A social exclusion paradigm ('cyberball' task) will be conducted post-training to evaluate VSOP training effects on social-emotional responses to social exclusion, including anxiety and motivation for social affiliation.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 60 years, community-dwelling, English-speaking, adequate vision and hearing for testing, capacity to give consent based on clinician assessment;
2. Telephone Interview for Cognitive Status (TICS) ≥ 31, Geriatric Depression Scale < 7 (i.e., free of major depression that can interfere with neural efficiency for social-emotional regulation), EXAMINER composite score (a comprehensive executive function battery test package that is sensitive to frontal regions' neural efficiency change) < .70 (i.e., reflecting decreased neural efficiency of frontal regions compared to cognitively health older adults in general);
3. moderate social relation difficulties: identified by World Health Organization Disability Assessment Scale (WHO-DAS), "Getting Along with Other People" domain, at least "moderate" difficulties endorsed; from HARP Database Project screening)

Exclusion Criteria:

1. a self-report clinical diagnosis of dementia or mild cognitive impairment;
2. MRI contraindications (e.g., pacemaker, metallic implant, claustrophobia);

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
cognitive capacity | baseline and 7 week post-training
  change of executive function from baseline to 7 week post-training

SECONDARY OUTCOMES:
brain function 1 (BOLD fMRI) | baseline and 7 week post-training
  brain functional change in response to social scenario task from baseline to 7 week post-training
social well-being | baseline and 7 week post-training
  change of social well-being measured by HARP Social Connectedness and Well-Being Core Battery from baseline to 7 week
brain function 2 (BOLD fMRI) | 7 week post-training only
  brain functional adaptability to cyberball task

CONTACTS AND LOCATIONS:
Overall Officials: Anne Corriveau, Study Director — University of Rochester
Locations (4):
- United States (4):
  - The Northfield, Fairport, New York
  - The Highlands, Pittsford, New York
  - River Edge Manor, Rochester, New York
  - St. Johns Meadows, Rochester, New York

IPD SHARING:
Plan to Share IPD: No